CLINICAL TRIAL: NCT06760299
Title: Investigation of the Effect of Kinesio Taping Applied to Lumbar Paravertebral Muscles Under Different Tensions on Local Body Temperature: a Single-Blind, Randomized Controlled Trial
Brief Title: Effect of Kinesio Taping on Lumbar Muscle Temperature
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Umut Ziya Kocak, Associate Professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1649B032404842; 1649B032404842 (Other Grant/Funding Number: TUBITAK (The Scientific and Technological Research Council of Türkiye) 2211-Graduate Scholarship Program)
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Kinesio Taping; Body Temperature Changes
Keywords: Thermal Imaging; Kinesio Taping; Body Temperature; Lumbar Muscles
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three groups: a 25% tension Kinesio Taping (KT) group, a 75% tension KT group, and a control group. Each group will receive a different intervention, with the KT applied unilaterally to the lumbar paravertebral muscles based on the designated tension level. The study is single-blind, meaning the researcher assessing the local body temperature using infrared thermography will be blinded to the group assignments. Temperature measurements will be taken at four time points: before the KT application, 15 minutes after, 45 minutes after, and 24 hours post-application, to assess the immediate and lasting effects of the KT interventions. The primary aim is to compare the impact of different KT tensions on local body temperature, serving as an indicator of changes in circulation and the therapeutic effect of KT.
Who Masked: Investigator
Masking Description: The participants will be aware of the group to which they are assigned (25% tension KT, 75% tension KT, or control group), but the researcher performing the thermal measurements using infrared thermography will be blinded to the group assignments. This ensures that the data collector's knowledge of the group assignment does not influence the measurement process or interpretation of the results. The masking of the researcher conducting the thermal imaging minimizes the risk of bias during data collection and analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 25% Tension Kinesio Taping Group (Active Comparator): Participants in this group will receive Kinesio Taping applied unilaterally to the lumbar paravertebral muscles with 25% tension. The tape will be applied using an "I" shaped strip with 5 cm anchor segments and 0% tension at both ends. The application will be conducted while the participant is in a neutral standing position, and the tape will be rubbed to ensure adhesion.
  Interventions: Other: %25 tension Kinesio tape
- Control Group (No Intervention): Participants in this group will not receive any Kinesio Taping intervention. This group will serve as a baseline for comparison with the KT groups, allowing for the assessment of the effects of KT on local body temperature.
- 75% Tension Kinesio Taping Group (Active Comparator): Participants in this group will receive Kinesio Taping applied unilaterally to the lumbar paravertebral muscles with 75% tension. The tape will be applied in an "I" shape with 5 cm anchor segments at both ends. The tension will be adjusted to 75% during the application, and the same adhesion process will be followed.
  Interventions: Other: 75% tension Kinesio tape

INTERVENTIONS:
Other: %25 tension Kinesio tape — "I" shaped Kinesio tape application with 25% tension
  Arms: 25% Tension Kinesio Taping Group
Other: 75% tension Kinesio tape — "I" shaped Kinesio tape application with 75% tension
  Arms: 75% Tension Kinesio Taping Group

SUMMARY:
This single-blind, randomized controlled trial aims to investigate the effect of Kinesio Taping (KT) applied to lumbar paravertebral muscles with different tensions (25% and 75%) on local body temperature. The study will compare the changes in local body temperature before and after KT application using infrared thermography. Participants will be randomly allocated to one of three groups with randomization stratified by sex: 25% tension KT, 75% tension KT, and a control group. Temperature measurements will be taken at four time points: before the application, 15 minutes, 45 minutes, and 24 hours post-application. The data will be analyzed using statistical methods to evaluate the impact of KT tension on local body temperature. This study will provide insights into the physiological effects of KT under different tension levels.

DETAILED DESCRIPTION:
This single-blind, randomized controlled trial aims to assess the effects of Kinesio Taping (KT) applied to the lumbar paravertebral muscles at different tension levels (25% and 75%) on local body temperature. KT is an elastic adhesive band that is believed to increase circulation, improve muscle function, support proprioception, and alleviate pain. Previous studies have explored the effects of KT on local temperature, but the impact of varying tension levels on temperature and circulation has not been extensively examined. This study seeks to fill this gap by investigating how different tensions in KT application affect local body temperature, a potential indicator of changes in circulation.

The study will include 54 participants, randomly assigned into three groups: a 25% tension KT group, a 75% tension KT group, and a control group. Participants will be stratified by gender to ensure balanced representation. KT will be applied unilaterally to the paravertebral muscles, with the side (right or left) selected by a coin toss. The KT application will follow the standard "I" shape, with 5 cm anchor segments at both ends, and the tension will be applied along the L1-L5 vertebrae in a neutral standing position. After participants bend forward to their maximum comfort level, the tape will be applied, and adhesion will be ensured by rubbing the tape.

Local body temperature will be measured using a FLIR E5 infrared camera (Teledyne FLIR, USA) at four time points: immediately before the KT application, 15 minutes after the application, 45 minutes after the application, and 24 hours post-application. The thermal measurements will be analyzed using FLIR E5 software to determine the minimum, average, and maximum temperatures of the taped area.

The primary outcome of the study is to determine if KT application under different tension levels influences local body temperature, potentially reflecting changes in blood circulation. Secondary outcomes include the comparison of temperature variations between the tension groups and the control group, and the analysis of how time influences these changes.

Statistical analysis will involve one-way analysis of variance (ANOVA) to compare the demographic characteristics of the groups and a three-way repeated measures ANOVA to assess differences in local body temperature across groups (25% tension, 75% tension, and control), sides (right and left), and time points. Bonferroni post hoc tests will be used to further explore significant interactions or main effects. Descriptive statistics will summarize demographic data, and significance will be set at p < 0.05.

This study is expected to provide valuable insights into the physiological effects of KT and may contribute to a better understanding of how different tension levels influence local circulation and body temperature. These findings could inform clinical practices related to KT and its potential therapeutic benefits.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study
* Aged between 18 and 35 years
* Ability to read and understand Turkish

Exclusion Criteria:

* Experiencing muscle pain in the upper extremity, torso, or lower extremity
* Use of medication or having a systemic disease that may affect thermoregulation
* Having dermatological conditions in the area where Kinesio Taping will be applied
* Having undergone surgery in the upper extremity, torso, or lower extremity
* Being pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Local Body Temperature | Temperature will be measured before, 15 minutes, 45 minutes, and 24 hours after KT removal using an infrared thermographic camera.
  The primary outcome measure of this study is the change in local body temperature in the lumbar paravertebral muscles following the application of Kinesio Taping (KT). Local body temperature will be measured using an infrared thermographic camera to assess the effect of KT on blood circulation and metabolic activity in the targeted area. The temperature measurements will focus on evaluating the difference in temperature at various time points after the application of KT.

SECONDARY OUTCOMES:
Thermal Data Analysis | Thermal data will be analyzed at the same time points as the primary outcome: immediately before Kinesio Taping application, 15 minutes after application, 45 minutes after application, and 24 hours after KT removal.
  The analysis of thermal data (minimum, average, and maximum temperatures) using FLIR software will support the primary measure but is considered secondary as it helps to further understand the impact of KT on circulation and tissue temperature.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi University Physiotherapy and Rehabilitation Research Laboratory, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
No consensus among researchers yet